CLINICAL TRIAL: NCT05377177
Title: Cortical Inhibition as a Biomarker of Response in a Comparison of Bilateral Versus Unilateral Accelerated Theta Burst Stimulation for Suicidal Ideation in Treatment-Resistant Depression (COMBAT-SI)
Brief Title: Cortical Inhibition as a Biomarker of Response in a Comparison of Bilateral Versus Unilateral Accelerated Theta Burst Stimulation for Suicidal Ideation in Treatment-Resistant Depression -COMBAT-SI
Acronym: COMBAT-SI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Cory Weissman, Medical Director of Interventional Psychiatry; Assistant Clinical Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 801566
Record Dates: First submitted 2022-03-24; First posted 2022-05-17 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Suicidal Ideation; Treatment-resistant Depression
Keywords: theta burst stimulation; accelerated TBS; bilateral TBS
MeSH Terms: conditions — Suicidal Ideation; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study will be randomized to bilateral vs. unilateral aiTBS in a 1:1 ratio . Treatments will be over 1 week.
Who Masked: Participant, Outcomes Assessor
Masking Description: A sham component will be used over the right DLPFC for unilateral aiTBS treatment. This treatment component will mitigate concerns of expectancy, and will lead to blinding for patients. The Cool B65 A/P coil is unmarked, with one side producing active treatment and the other sham treatment with concurrent electrical stimulation, which accurately mimics active stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bilateral aTBS (Experimental): Patients will receive Bilateral accelerated theta-burst stimulation bilaterally for 5 consecutive days, with a total of 10 hours a day. treatment will be 10min with 50min of breaks in between the 10 sessions.
  Interventions: Device: Accelerated Theta Burst Stimulation
- Unilateral aiTBS (Active Comparator): Patients will receive unilateral accelerated theta-burst stimulation to the left side for 5 consecutive days, with a total of 10 hours a day. treatment will be 10min with 50min of breaks in between the 10 sessions. There will be a right DLPFC sham component to this treatment arm for all treatment sessions.
  Interventions: Device: Accelerated Theta Burst Stimulation

INTERVENTIONS:
Device: Accelerated Theta Burst Stimulation — B65 magnetic coil stimulation applied to the dorsal lateral prefrontal cortex.

SUMMARY:
This is a prospective clinical trial to confirm the effectiveness of bilateral accelerated theta burst stimulation (aTBS) on suicidal ideation (SI), while exploring cortical inhibition measures in this treatment paradigm. In this proposed study, the investigators will evaluate the anti-suicidal effects of bilateral aTBS over the DLPFC compared to accelerated intermittent theta burst stimulation (aiTBS) over the left DLPFC in participants with TRD and SI. Additionally, the investigators aim to identify neurophysiological targets through which bilateral aTBS induces remission of SI in TRD differentially from aiTBS.

DETAILED DESCRIPTION:
Suicidality is a growing epidemic, as over 700,000 people die by suicide around the world annually. Current treatments for suicidality are limited and novel treatments for suicidality are desperately needed. There is early evidence to suggest that the non-invasive brain stimulation treatment called repetitive transcranial magnetic stimulation, or rTMS, is better than placebo at eliminating suicidal ideation (SI) in patients with hard to treat depressive illness (treatment-resistant depression; TRD). The UCSD Interventional Psychiatry lab was the first group to demonstrate that bilateral rTMS, targeted to specific areas of the frontal lobes of the brain, is more effective than placebo for SI. Recent evidence from the lab also showed that improvement in SI with brain stimulation treatment is correlated with changes in specific measures of neuronal communication, that is cortical inhibition, in these same brain regions. A prospective clinical trial to confirm the effectiveness of bilateral rTMS on SI, while exploring cortical inhibition measures in this treatment paradigm, is prudent and urgently needed. In this proposed study, the investigators plan to evaluate the anti-suicidal effects of bilateral aTBS over the DLPFC (an accelerated form of rTMS delivered with multiple theta burst treatments per day) compared to aiTBS over the left DLPFC in participants with TRD and SI. Additionally, the investigators aim to identify neurophysiological targets through which bilateral aTBS induces remission of SI in TRD differentially from aiTBS.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old.
2. Diagnosis of major depressive episode, confirmed on Mini-International Neuropsychiatric Interview (MINI), with HRSD score ≥18.
3. Ongoing SI present beyond screening phase of study (confirmed with Beck SSI score ≥4).
4. Pass the TMS adult safety screening (TASS) questionnaire and the MRI safety screening questionnaire.
5. Have failed to achieve a clinical response to an adequate dose of two antidepressants based on an Antidepressant Treatment History Form (ATHF) score for each antidepressant trial of > 3 in the current episode OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF score of 1 or 2 on those 2 separate antidepressants) OR have a combination of one failed trial and one not tolerated trial, per the definitions above.
6. Psychiatric illness due to a general medical condition (GMC) has been ruled out during initial assessment.
7. Voluntary outpatients capable to consent to treatment and seen at the UC San Diego Health Interventional Psychiatry program.
8. Able to adhere to the treatment schedule.

Exclusion Criteria:

1. Have a confirmed diagnosis of substance use disorder within the last 3 months.
2. Have a lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms.
3. Have a diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, that is assessed by a study investigator to be primary and causing greater impairment than MDD.
4. Have a diagnosis of any personality disorder, and assessed by a study investigator to be primary and causing greater impairment than MDD.
5. Have SI prompting emergent involuntary hospital stay (SI in which the participant can maintain voluntary and capable outpatient status as well as recent suicide attempt will not be exclusionary).
6. Currently pregnant or lactating, or woman or childbearing age without adequate birth control.
7. Non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).
8. Not capable to consent to treatment and/or not suitable for outpatient treatment.
9. Have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump; Have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT or a febrile seizure of infancy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than 5 minutes; Have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
10. Currently take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in scores on the suicide scale index (SSI) from baseline | 6-months
  The primary outcome will be a comparison of change in score on the suicidality scale index (SSI) from baseline to endpoint of treatment between accelerated bilateral and unilateral treatment. The SSI contains 19 items scored from 0 to 2, higher scores indicating more severity, with overall scores ranging from 0 to 38The primary endpoint will be at treatment completion for both arms. The investigators will follow patients at 1, 2, 3, and 4 weeks post-treatment, as well as 3 and 6 months after treatment completion.

SECONDARY OUTCOMES:
Neurophysiological measures of cortical inhibition, N100, short interval cortical inhibition, and cortical evoked activity | 6-months
  Analysis of transcranial magnetic stimulation concurrent with electroencephalogram (TMS-EEG) to extract effective connectivity metrics between the subgenual cingulate (SGC) and the dorsolateral prefrontal cortex (DLPFC) as suicidality biomarkers, as measured by changes in scores on the SSI, for left aiTBS compared to bilateral aTBS.
Categorical suicidal clinical outcomes | 6-months
  Suicide attempts and completions will be recorded as adverse events throughout the duration of the study. The investigators will complete categorical sensitivity analyses for these outcomes between treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Interventional Psychiatry, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT05377177/Prot_ICF_000.pdf